CLINICAL TRIAL: NCT01133873
Title: A Randomized, Multiple-Dose, Double-Blind, Placebo-Controlled Study of Sequential Ascending Dose Levels to Assess the Safety, Tolerability and Electrocardiographic Effects of Propoxyphene Napsylate Capsules (and Its Metabolite Norpropoxyphene) When Administered Orally to Healthy Adult Subjects
Brief Title: Multiple-Ascending-Dose Study to Evaluate the Safety of Propoxyphene Napsylate In Healthy Adult Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Xanodyne Pharmaceuticals (Industry)
Responsible Party: Gary Shangold, MD / Chief Medical Officer, Xanodyne Pharmaceuticals, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: XP20C-101
Record Dates: First submitted 2010-05-24; First posted 2010-05-31 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
MeSH Terms: interventions — propoxyphene napsylate; Levopropoxyphene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Propoxyphene napsylate (XP20C)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propoxyphene napsylate (XP20C) — 100 mg capsules 6 times a day in ascending doses until a maximum tolerated dose is identified
  Other Names: propoxyphene napsylate; Darvon-N; XP20C
  Arms: 1
Drug: Placebo — 6 times a day in ascending doses until a maximum tolerated dose is identified
  Arms: 2

SUMMARY:
The purpose of this study is to determine the daily maximum tolerated dose of propoxyphene napsylate in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 18 and ≤ 30 (kg/m2)
* Medically healthy with normal screening results, or in the case of results that are abnormal; the abnormal results are clinically insignificant (eg, medical history, physical examination, neurological assessment, vital signs, oxygen saturation, laboratory profiles)
* 12-lead ECGs (calculations by the electrocardiograph) which have no clinically significant findings
* Vital signs which are within normal range
* No tobacco/nicotine-containing product use for a minimum of 6 months
* If female, must be able to adhere to acceptable methods of contraception or be postmenopausal or surgically sterile

Exclusion Criteria:

* History or presence of significant cardiovascular, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, or neurological disease
* History or presence of any degree of chronic obstructive pulmonary disease
* History of suicidal ideations or depression requiring professional intervention including counseling or antidepressant medication
* Any history of drug or alcohol abuse
* Positive drug (urine)/alcohol (breath) testing at screening or check-in
* Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV)
* History of hypersensitivity or allergy to propoxyphene or any opioid compound, naloxone, naltrexone, palonosetron (Aloxi®), glycerin, senna, or bisacodyl (Dulcolax®)
* Use of any prescription medication (with the exception of hormonal contraceptives for females) within 2 weeks of enrollment
* Use of any over-the-counter medication, including herbal products, within 1 week of enrollment
* Use of any drugs known to significantly inhibit or induce liver enzymes involved in drug metabolism [CYP P450]) within 30 days of enrollment
* Blood donation or significant blood loss within 30 days of enrollment
* Plasma donation within 7 days of enrollment
* Participation in another clinical trial within 30 days of enrollment
* Females who are pregnant or lactating
* Any other condition or prior therapy, which, in the opinion of the PI, would make the subject unsuitable for this study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of propoxyphene napsylate as determined by evaluation of adverse events, change from baseline of ventricular repolarization, lab results, and mental status | Day 13

SECONDARY OUTCOMES:
Establish the relationship between serum concentrations of propoxyphene and norpropoxyphene on cardiac conduction and pharmacokinetic linearity of sequentially increased dose levels of propoxyphene napsylate. | Days -1, 1, 4, 11

CONTACTS AND LOCATIONS:
Overall Officials: Lynn R Webster, MD, Principal Investigator — Lifetree Clinical Research
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States